CLINICAL TRIAL: NCT06879899
Title: MRD-Guided Surveillance in Locally Advanced Mid-Low Rectal Cancer (SURVEILLANCE-III)
Acronym: SURIII
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Director of Colorectal Surgery Department, Zhongshan hospital, Fudan University, Fudan University
Other Study IDs: SURVEILLANCE-III
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — In this study, the specific types of samples that will be retained are peripheral blood samples collected from patients at multiple time points. These samples will be used for circulating tumor DNA (ctDNA) analysis to assess minimal residual disease (MRD) status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MRD-Guided Surveillance in Locally Advanced Mid-Low Rectal Cancer

SUMMARY:
This study aims to explore the relationship between minimal residual disease (MRD) status and disease recurrence in patients with locally advanced mid-low rectal cancer. MRD refers to the presence of cancer cells that remain in the body after treatment but are undetectable by traditional imaging methods. The study will use a blood-based circulating tumor DNA (ctDNA) methylation test to assess its ability to predict cancer recurrence and survival outcomes.

Patients who are newly diagnosed with cT3/N+, M0 mid-low rectal cancer (tumor ≤10 cm from the anal verge) and are eligible for curative-intent treatment will be enrolled. Blood samples will be collected at multiple time points, including before neoadjuvant therapy, before surgery, after surgery, and during follow-up visits over three years. The study will compare MRD status with disease-free survival (DFS), recurrence-free survival (RFS), overall survival (OS), and the time it takes for MRD to detect recurrence compared to standard imaging methods.

The goal is to determine whether MRD monitoring can provide an early warning of cancer recurrence and help guide treatment decisions. This study may offer valuable insights into improving postoperative surveillance and personalized treatment strategies for rectal cancer patients.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study designed to evaluate the effectiveness of ctDNA-based MRD monitoring in predicting disease recurrence and survival outcomes in patients with locally advanced mid-low rectal cancer. The study will enroll 139 patients who have not previously received chemotherapy, radiotherapy, or targeted therapy.

Key Objectives

Primary Objective:

To explore the correlation between MRD status and disease-free survival (DFS) in locally advanced mid-low rectal cancer patients.

Secondary Objectives:

To assess the relationship between MRD status and 1-year/2-year recurrence-free survival (1yRFS, 2yRFS).

To evaluate the association between MRD status and overall survival (OS).

Exploratory Objectives:

To determine the average time by which MRD detection precedes imaging-based detection of disease recurrence.

To assess the correlation between post-neoadjuvant therapy MRD status and pathological complete response (pCR).

Study Design

Patients will undergo blood sampling at key time points:

Baseline (pre-neoadjuvant therapy) Pre-surgery (0-7 days before surgery) Post-surgery (7±2 days after surgery) Follow-up visits at 1, 3, 6, 9, 12, 18, 24, and 36 months post-surgery MRD status will be assessed using a ctDNA methylation-based PCR test, which provides a rapid, cost-effective alternative to traditional NGS-based methods.

Statistical Analysis Kaplan-Meier survival analysis will be used to estimate DFS, RFS, and OS. Cox proportional hazards models will assess whether MRD status serves as an independent prognostic factor for recurrence.

Multivariate analysis will adjust for clinical variables, including tumor burden and treatment history.

Ethical Considerations The study adheres to the principles of the Declaration of Helsinki and Chinese Good Clinical Practice (GCP) guidelines.

Informed consent will be obtained from all participants, and privacy and confidentiality will be strictly maintained.

Expected Outcomes This study aims to validate the clinical utility of ctDNA-based MRD monitoring in predicting recurrence and survival outcomes for locally advanced mid-low rectal cancer patients. If successful, MRD testing may offer a more effective tool for postoperative surveillance and treatment planning, allowing for earlier interventions and improved long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1） Age 18-80 years old, male or female; 2) histologically confirmed diagnosis of rectal adenocarcinoma (i.e., adenoepithelial carcinoma, including adenocarcinoma, mucinous carcinoma, imprinted cell carcinoma, and undifferentiated carcinoma; excluding adenosquamous carcinoma); 3) Preoperative clinical stage cT3 /N+, M0, the lower edge of the tumor is ≤10cm from the anal verge, and no surgical resection is performed; (4) Not receiving chemotherapy, radiotherapy, targeted therapy or other anti-tumor therapy; 5) Radical surgery is available; 6) ECOG score 0-1; 7) Subjects voluntarily enrolled in this study and signed the informed consent, good compliance, follow the planned schedule and actively cooperate with the return to the hospital for regular clinical follow-up and necessary treatment.

Exclusion Criteria:

1. previous other malignant tumors (including non-adenocarcinoma colorectal cancer);
2. Previously received other anti-tumor therapy;
3. Pregnant and lactating women; (4) Patients with other medical conditions that, in the judgment of the investigator, may interfere with follow-up and short-term survival;

5) Subjects have other factors that may lead to forced termination of this study, such as other serious illnesses (including mental illness, infectious diseases, fever ≥38℃, etc.) that require combined treatment, serious laboratory test abnormalities, accompanied by family or social factors that will affect the safety of the subjects, or the collection of data and samples.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with locally advanced mid-low rectal cancer (cT3/N+, M0, tumor ≤10 cm from the anal verge) who have not received prior treatment. Participants will be recruited from multiple clinical centers and must meet specific eligibility criteria to ensure the study's validity.
  Key Characteristics of the Study Population:
  Diagnosis: Histologically confirmed rectal adenocarcinoma (including adenocarcinoma, mucinous adenocarcinoma, signet-ring cell carcinoma, and undifferentiated carcinoma; excluding adenosquamous carcinoma).
  Stage: Clinical locally advanced mid-low rectal cancer (cT3/N+, M0) confirmed by preoperative imaging and clinical assessment.
  Treatment History: No prior chemotherapy, radiotherapy, targeted therapy, or other anti-cancer treatments.
  Surgical Eligibility: Candidates must be eligible for curative-intent surgery following neoadjuvant therapy.
  General Health Status: ECOG performance status 0-1, indicating good functional status
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Exploring the correlation between MRD status and disease-free survival (DFS) in patients with locally progressive low and intermediate rectal cancer | From surgery to disease recurrence or up to 36 months
  Exploring the correlation between MRD status and disease-free survival (DFS) in patients with locally progressive low and intermediate rectal cancer

SECONDARY OUTCOMES:
Correlation of MRD status with 1-year recurrence-free survival (1yRFS) | From surgery to 12 months
  Correlation of MRD status with 1-year recurrence-free survival (1yRFS)
Correlation of MRD status with 2-year event-free survival (2yRFS) | From surgery to 24 months
  Correlation of MRD status with 2-year event-free survival (2yRFS)
Correlation of MRD status with overall survival (OS) | From surgery to death or up to 36 months
  Correlation of MRD status with overall survival (OS)

OTHER OUTCOMES:
MRD detects disease recurrence earlier than imaging (CT) average advance time | From surgery to disease recurrence, assessed up to 36 months
  MRD detects disease recurrence earlier than imaging (CT) average advance time
Correlation between MRD status and pathologic complete remission rate (pCR) after neoadjuvant therapy | From completion of neoadjuvant therapy to surgery
  Correlation between MRD status and pathologic complete remission rate (pCR) after neoadjuvant therapy

IPD SHARING:
Plan to Share IPD: No